CLINICAL TRIAL: NCT07252752
Title: Dopamine and Insulin in Psychosis: Imaging the Effects of Intranasal Insulin on Dopamine Transmission
Brief Title: Dopamine and Insulin in Psychosis
Acronym: DIPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Matthäus Willeit, Ao. Univ. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: KLP4656125
Record Dates: First submitted 2025-09-30; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: First Episode Psychosis (FEP)
Keywords: positron emission tomography (PET); dopamine; schizophrenia; intranasal insulin; magnetic resonance spectroscopy (MRS)
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Schizophrenia group (Experimental): 20 antipsychotic-naive patients with first episode psychosis will undergo (i) two [11C]-(+)-PHNO PET scans preceded by intranasal insulin or placebo administration in a randomized counterbalanced order, and (ii) 1H-MRS before and after intranasal insulin
  Interventions: Drug: Intranasal Insulin; Drug: Placebo; Drug: Low dose insulin infusion; Drug: Placebo infusion; Radiation: [11C] (+)-4-propyl-(+)-4-propyl-9-hydroxynaphthoxazine (PHNO)
- Healthy volunteer group (Experimental): 20 healthy volunteers will undergo (i) two [11C]-(+)-PHNO PET scans preceded by intranasal insulin or placebo administration in a randomized counterbalanced order, and (ii) 1H-MRS before and after intranasal insulin
  Interventions: Drug: Intranasal Insulin; Drug: Placebo; Drug: Low dose insulin infusion; Drug: Placebo infusion; Radiation: [11C] (+)-4-propyl-(+)-4-propyl-9-hydroxynaphthoxazine (PHNO)
- Test-retest group (Other): 6 healthy volunteers will undergo (i) two [11C]-(+)-PHNO PET scans, and (ii) 1H-MRS for test-retest purposes
  Interventions: Radiation: [11C] (+)-4-propyl-(+)-4-propyl-9-hydroxynaphthoxazine (PHNO)

INTERVENTIONS:
Drug: Intranasal Insulin — 160 IU intranasal insulin is administered using precision air pumps twice: 15 min prior to the PET scan and 35 min prior to the 1H-MRS scan
  Arms: Healthy volunteer group; Schizophrenia group
Drug: Placebo — Insulin-free dilution buffer is administered using precision air pumps 15 min prior to the PET scan
  Arms: Healthy volunteer group; Schizophrenia group
Drug: Low dose insulin infusion — 2.5 mU/kg insulin in 100 ml isotonic saline is infused intravenously over 15min prior to PET scan when placebo is administered intranasally
  Arms: Healthy volunteer group; Schizophrenia group
Drug: Placebo infusion — 100 ml saline is infused intravenously over 15min prior to PET scan when insulin is administered intranasally
  Arms: Healthy volunteer group; Schizophrenia group
Radiation: [11C] (+)-4-propyl-(+)-4-propyl-9-hydroxynaphthoxazine (PHNO) — Each participant undergoes a 90-min [11C]-(+)-PHNO scan twice

SUMMARY:
Patients with schizophrenia have a high risk of developing metabolic disorders and current evidence points to an overlap in mechanisms underlying psychiatric symptoms and metabolic disturbances. The main goal of this study is to investigate effects of brain insulin on dopamine signaling and energy metabolism in patients with schizophrenia experiencing their first psychotic episode (FEP). To this end, patients with schizophrenia and healthy volunteers will undergo two [11C]-(+)-PHNO positron emission (PET) scans to measure the changes in dopamine receptor availability after nasally applied insulin, as well as single proton magnetic resonance spectroscopy (1H-MRS) to assess the impact of intranasal insulin on levels of glucose and glutamate in the hippocampus.

ELIGIBILITY:
Inclusion Criteria:

All participants

* age 18-40
* Body mass index (BMI) range 18-25
* good general health according to physical examination and medical history
* absence of relevant abnormalities in laboratory screening, electrocardiogram (ECG) or vital signs
* no regular use of drugs of abuse or alcohol based on history and urine drug screen

Patients only

* diagnosis of schizophrenia or schizophreniform disorder according to DSM-5
* ability to give informed consent
* minimum Positive and Negative Syndrome Scale (PANSS) score of 55 with >3 on at least two or >4 on one PANSS psychosis item

Exclusion Criteria:

All participants

* severe or unstable medical or neurological illness or clinically significant abnormality on screening laboratory studies or ECG
* established diagnosis of type 1 or type 2 diabetes
* current substance use disorder or regular recreational drug abuse (except nicotine and caffeine)
* pregnancy or breastfeeding
* history of head trauma resulting in loss of consciousness of >1min or requiring medical attention
* presence of MRI exclusion criteria
* if participation in this study would exceed annual radiation dose limits (30mSv)
* clinically established diagnosis of intellectual disability

Healthy volunteers only

* Psychiatric disorder according to Mini-International Neuropsychiatric Interview (M.I.N.I.)
* Schizophrenia or bipolar disorder in first degree family members

Patients only

● Previous oral antipsychotic treatment for more than 2 weeks or previous treatment with antipsychotic depot preparation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
[11C]-(+)-PHNO BPND values | Assessed on two separate study visits within 5-12 days (scan duration: 90 min)
  Dopamine D2/3 receptor availability after intranasal insulin or placebo administration
Hippocampal glucose and glutamate concentrations | Assessed during a single study visit (scan duration: 40 min in total)
  Hippocampal glucose and glutamate concentrations before and after intranasal insulin administration

SECONDARY OUTCOMES:
Changes in blood-based parameters of energy metabolism | Assessed at baseline and at 15min intervals after instranasal insulin/placebo administration over a period of up to 90min
  Changes in concentrations of selected metabolic parameters (blood glucose, insulin, c-peptide, total cholesterol, HDL, LDL, trigycerides, ketone bodies) following intranasal insulin/placebo administration, assessed by venous blood sampling
Hippocampal volumetric parameters | Assessed during a single study visit, at baseline (scan duration: 10min)
  Whole hippocampus and hippocampal subfield volumes assessed with structural MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided